CLINICAL TRIAL: NCT02498561
Title: Phase 1 Study of Periodontal Disease and Obese Individuals That Investigate of Local and Systemic Antioxidant Levels of Before and After Periodontal Treatment
Brief Title: The Effects of Obesity on Glutathione Levels in Patients With Chronic Periodontitis Before and After Periodontal Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Figen ÖNGÖZ DEDE (Other)
Collaborators: Bulent Ecevit University (Other)
Responsible Party: Sponsor-Investigator, Figen ÖNGÖZ DEDE, Faculty of Dentistry, Bulent Ecevit University
Organization: Bulent Ecevit University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 2013-62550515-02
Record Dates: First submitted 2015-07-09; First posted 2015-07-15 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- obese-chronic periodontitis patients (Active Comparator): GCF, plasma and GCF samples were taken before and after nonsurgical periodontal therapy
  Interventions: Procedure: nonsurgical periodontal therapy
- obese-periodontally healthy controls (Placebo Comparator): GCF, plasma and GCF samples were taken at baseline after oral hygiene instructions
  Interventions: Procedure: oral hygiene instructions
- normal weight-CP patients (Active Comparator): GCF, plasma and GCF samples were taken before and after nonsurgical periodontal therapy
  Interventions: Procedure: nonsurgical periodontal therapy
- normal weight-PH controls (Placebo Comparator): GCF, plasma and GCF samples were taken at baseline after oral hygiene instructions
  Interventions: Procedure: oral hygiene instructions

INTERVENTIONS:
Procedure: nonsurgical periodontal therapy — Scaling and root planning under local anaesthesia, in a total of four clinical visits Oral hygiene instructions including the modified Bass technique, regular toothpaste, and an appropriate interdental cleaning device with dental floss and interdental brush.
  Other Names: obese-chronic periodontitis patients
  Arms: obese-chronic periodontitis patients
Procedure: oral hygiene instructions — Oral hygiene instructions including the modified Bass technique, regular toothpaste, and an appropriate interdental cleaning device with dental floss and interdental brush
  Other Names: obese-periodontally healthy controls
  Arms: obese-periodontally healthy controls
Procedure: nonsurgical periodontal therapy — Scaling and root planning under local anaesthesia, in a total of four clinical visits Oral hygiene instructions including the modified Bass technique, regular toothpaste, and an appropriate interdental cleaning device with dental floss and interdental brush.
  Other Names: normal weight-CP patients
  Arms: normal weight-CP patients
Procedure: oral hygiene instructions — Oral hygiene instructions including the modified Bass technique, regular toothpaste, and an appropriate interdental cleaning device with dental floss and interdental brush
  Other Names: normal weight-PH patients
  Arms: normal weight-PH controls

SUMMARY:
Obesity may affect periodontal health by inducing gingival oxidative damage through increased production in circulating reactive oxygen species (ROS). Previous studies have reported decreased glutathione levels in patients with periodontitis when compared to healthy subjects in gingival crevicular fluid (GCF), plasma and saliva. In the present study we hypothesized that high ROS levels in circulation may decrease glutathione levels in the GCF,plasma and saliva in obese patients with chronic periodontitis, whereas periodontal therapy could have positive effects on glutathione levels.

DETAILED DESCRIPTION:
The purpose of this study was to investigate the effects of obesity on glutathione levels in the plasma, GCF and saliva of patients with chronic periodontitis and to evaluate changes after nonsurgical periodontal therapy.

Diagnosed as obese (n=30) and normal-weight (n=30) individuals were categorized; chronic periodontitis (CP) and periodontally healthy controls (PH). Gingival crevicular fluid (GCF), plasma, saliva samples and clinical measurements were obtained at baseline and a month after nonsurgical periodontal therapy.

Unstimulated salivary samples were collected using standard techniques. About 2 mL whole saliva was collected in disposable tubes and centrifuged immediately to remove cell debris (10,000 g x 10 minutes). The supernatants (50µL each) were stored at -40C until analyzed. GCF samples were collected from a mesio-buccal and disto-palatal site on each tooth. In the CP group, the samples were obtained from patients at areas with ≥5 mm CAL, ≥6 mm PD and ≥30% bone loss. In gingivitis group, GCF samples were obtained from teeth with BOP and without CAL. In the healthy group, GCF samples were collected from teeth exhibiting PD<3 mm without CAL and BOP. The area was isolated with cotton rolls, saliva contamination elimination was ensured, and it was slightly air dried. GCF was sampled with paper strips. Paper strips were placed into the crevice until mild resistance was felt (intracrevicular method) and left in the position for 30 seconds. Strips contaminated with blood or saliva were discarded. Each sampled strip was placed into a 400µl eppendorf centrifuge tube and stored at -40C until analyzed.

Five milliliters of venous blood was taken from antecubital vein by using a standard venipuncture method. Obtained blood sample was collected in vacutainer tubes and anti-coagulated with EDTA. The blood samples were then stored at -40C until required for use in ELISAs.

Power analysis indicated that 12 individuals for each group would be sufficient to achieve 80% power to detect a difference of 0.05 between the alternative and the null hypotheses.

The Shapiro Wilk test was used to investigate whether or not the data were normally distributed. Continuous variables with unequal variances were compared by means of Welch and Tamhane's T2 post-hoc test for BMI, PD, CAL and the levels of glutathione. The comparison of the age, GI, PI and BOP was analyzed using the Kruskal-Wallis non-parametric test followed by post hoc group comparisons with the Bonferroni-adjusted Mann-Whitney U test. Paired Student's t-test or Wilcoxon rank-sum test was used to compare the measurements at two points (baseline and after SRP). The Spearman's rank correlation test was also used to detect the relationship between biochemical and clinical findings.

ELIGIBILITY:
Inclusion Criteria:

* never-smokers
* no history of systemic disease
* no patients had been under periodontal therapy and medicine for at least 6 months before the study
* no pregnancy or lactation
* no alcohol or antioxidant vitamin consumption.

Exclusion Criteria:

-

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-03; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Biochemical parameters (GSH and GSSG levels, GSH/GSSG ratio ) | Baseline and 1 month after treatment
  The changes in levels of reduced and oxidized glutathione (GSH and GSSG) 1 month after periodontal treatment determined by ELISA. The changes in levels of GSH were analyzed to determine diagnostic and prognostic potential as a biomarker of periodontitis and obesity.

SECONDARY OUTCOMES:
Probing pocket depth | Baseline and 1 month after treatment
  The changes in probing pocket depth after periodontal treatment.Probing pocket depth was measured for determining severity of disease and clinic outcome.
Probing pocket depth and clinical attachment level | Baseline and 1 month after treatment
  The changes in clinical attachment level after periodontal treatment. The probing depth and the distance from the gingival margin to the cemento-enamel junction are used to measurement of clinical attachment level. Clinical attachment level was measured for determining severity of disease and clinic outcome.
Gingival index | Baseline and 1 month after treatment
  he changes in gingival index after periodontal treatment. Gingival index was recorded for classifying and evaluating (coronally) gingival inflammation.
Plaque index | Baseline and 1 month after treatment
  The changes in plaque index after periodontal treatment. Plaque index was recorded for determining and classifying oral hygiene status.
Bleeding on probing | Baseline and 1 month after treatment
  The changes in bleeding on probing after periodontal treatment. Bleeding on probing was recorded for classifying and evaluating (apically) gingival inflammation.